CLINICAL TRIAL: NCT05276349
Title: Home-based Remote Digital Monitoring to Assess ALS Progression (Track ALS)
Status: Completed | Type: Observational
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Emory University (Other); Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DHI-10012021-ALS
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to study use of advance Digital Health Technologies (DHT) and its validity as measures for assessing progression in Amyotrophic Lateral Sclerosis (ALS) patients. A total of 80 ALS patients will be recruited across US, and will involve two sites - St. Joseph Hospital and Medical Center in Phoenix, AZ, and Emory University ALS Clinic in Atlanta. This will be a fully remote observational study and will employ remote data collection platforms such as (a) A digital spirometry device powered by a mobile app will be used to measure vital capacity; (b) A clinical-grade voice recording app will be used to evaluate speech function; (c) A medical-grade wearable sensor will be used to monitor activity levels and sleep patterns; and (d) Standardized Electronic Clinical Outcome Assessments (eCOA) and Patient Reported Outcomes (ePRO) will be used to evaluate quality of life and cognitive abilities.

The main goals of this study is to answer some of these questions:

1. Can ALS patients measure important aspects of disease progression at home, either by themselves with appropriate training or with assistance of a coordinators via virtual visit?
2. Which clinical outcome measures collected through DHT are sensitive indicators of ALS progression?
3. Are the measures reproducible and whether they can correlate with gold standard assessments?

The results of this study have the potential to provide valuable information for designing future ALS trials that are more decentralized, more patient-centric, and require less visits to the clinic which typically become a major burden with disease progression

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 90.
2. Diagnosed with definite, probable, or possible ALS according to the modified El Escorial Criteria (EEC) or diagnosed with ALS using the Gold Coast Criteria.
3. Must be able to ambulate independently at the time of enrollment, with or without the use of foot braces or cane.
4. A vital capacity score of ≥40% of the predicted value (at last known in-person visit and if available).
5. Intelligible speech with occasional repetition.
6. Willingness and medical ability to comply with scheduled visits and study procedures.
7. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI).
8. Possession of a smartphone, and willingness to install study apps on it.
9. Continuous internet access at home, with stable broadband internet access.
10. Sufficiently proficient in English to understand and complete questionnaires and follow instructions using smartphone apps.

Exclusion Criteria:

1. Diagnosed with a superimposed medical condition that could confound study procedures in the opinion of the investigator.
2. Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the participant's ability to comply with the protocol.
3. Any other reasons that, in the opinion of the PI, the candidate is determined to be unsuitable for entry into the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the ALS patient populations cared for at the BNI and Emory University ALS Clinics. For the virtual recruitment of ALS patients outside of those clinics, the study details with contact information will be posted on IRB-approved websites, social media, and patient advocacy groups, including the Northeast ALS Consortium (NEALS), ALS Association (ALSA) websites and other ALS forums. The National ALS Registry will also be used to promote recruitment.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of at-home assessments | 12 months
  The average number of at-home assessments completed by each subject will be calculated each quarter using Wald method

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No